CLINICAL TRIAL: NCT00651066
Title: Pharmacokinetics of Rifabutin Combined With Antiretroviral Therapy in the Treatment of Tuberculosis Patient With HIV Infection in Vietnam : A Phase II Trial
Brief Title: Pharmacokinetics of Rifabutin Combined With Antiretroviral Therapy in Patients With TB/HIV Co-infection in Vietnam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANRS12150b
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; Tuberculosis; Rifabutin; Pharmacokinetics; Vietnam
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): RBT (150 mg TPW during 3 weeks switch to 150mg OD for the following 3 weeks) associated with LPV/r based ART
  Interventions: Drug: rifabutin in combination with lopinavir boosted by ritonavir - dosing schedule 1
- 2 (Experimental): RBT (150 mg OD during 3 weeks switch to 150mg TPW for the following 3 weeks) associated with LPV/r based ART
  Interventions: Drug: rifabutin in combination with lopinavir boosted by ritonavir - dosing schedule 2

INTERVENTIONS:
Drug: rifabutin in combination with lopinavir boosted by ritonavir - dosing schedule 1 — 3TC(300mg)/D4t(60mg)/LPV/r(800mg/200mg)+INH/PZA/EMT/Rifabutin(150 mg TPW 3 wks switch to 150 mg OD 4 wks);
  Arms: 1
Drug: rifabutin in combination with lopinavir boosted by ritonavir - dosing schedule 2 — 3TC(300mg)/D4t(60mg)/LPV/r(800mg/200mg)+INH/PZA/EMT/Rifabutin(150 mg OD 3 wks switch to 150 mg TPW 4 wks);
  Arms: 2

SUMMARY:
The overall aim of the project is to evaluate rifabutin (RBT) as a replacement for rifampicin (RMP), for the combined treatment of tuberculosis and HIV infection. RBT represents an alternative to RMP for HIV infected patients as its half-life is longer and the enzymatic induction effect appears to be less important on the associated antiretroviral therapy (ART) drugs.

This phase II trial is to determine precisely the pharmacokinetics parameters of RBT in combination with different ART regimens in Vietnamese HIV infected patients with pulmonary tuberculosis, in order to define optimal doses that will be further tested in a larger phase III trial comparing safety, tolerability and efficacy of RBT and RMP regimens.

DETAILED DESCRIPTION:
Patients will be offered to participated in the study when they start TB treatment. All the enrolled patients will immediately be switched to rifabutin and randomized, to one of the RBT doses that will be then adapted to the allocated RBT regimen according to a cross over scheme. Three full pharmacokinetics profile will be performed at different time point : before initiation of ARV, after three weeks of the first RBT dosage and after three weeks of the secondRBT dosage. Patients will then be referred to the national program for further treatment. A follow-up visit will be planned at the end of the antiTB treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary tuberculosis defined as either

  * at least 2 sputum smears positive for AFB
  * 1 sputum smear positive for AFB and a chest radiograph compatible with active tuberculosis
  * 1 sputum culture positive and and a chest radiograph compatible with active tuberculosis
  * a clinical history and chest radiograph compatible with active tuberculosis and 2 sputum smear negative for AFB
* Positive HIV antibody and CD4 count <=250 /mm3
* Weight > 40 kg
* No history of ART
* No grade 3 or 4 clinical or laboratory findings
* Negative pregnancy test and appropriate contraceptive measures during the duration of the trial for female of childbearing age
* Having a firm home address that is readily accessible
* Karnofsky score>=80%

Exclusion Criteria:

* History of TB or MDR TB treatment
* Concomitant OI requiring additional anti-infectious treatment
* Formal contraindication to any drug used in the trial
* Diabetes mellitus requiring drug treatment
* Recreational drug or alcohol abuse
* History of drug hypersensitivity to TB or related medications
* Interrupted TB therapy for more than 1 week
* Less than 90% adherent to first 6 weeks of intensive phase chemotherapy
* Mental illness that could impair ability to give informed consent or result in poor adherence to trial protocol and therapy
* Neutropenia <1200 /L, anaemia <6.8 g/dL, liver function test > grade 2
* Requiring concomitant medications that may potentially interact with study drugs
* Pregnant or lactating women
* Karnofsky score >80%
* Any condition rendering the patient unable to understand the nature, scope, and possible consequences of thes study and to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of rifabutine measured (a)before introduction of ART;(b)after ART initiation (two different doses of RBT in combination with lopinavir/ritonavir) | 2, 5 and 8 weeks after randomisation

SECONDARY OUTCOMES:
Area under the curve (AUC) of lopinavir/ritonavir in combination with two doses of rifabutine | 5 and 8 weeks after randomisation
Safety : proportion of patients with grade 3 and grade 4 adverse events | through out the trial

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D. Harries, PhD, Principal Investigator — The international Union Against Tuberculosis and Lung Diseases (IUATLD), Paris, France; Huy Dung Nguyen, MD, Principal Investigator — Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam
Locations (1):
- Pham Ngoc Tach Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Lan NT, Thu NT, Barrail-Tran A, Duc NH, Lan NN, Laureillard D, Lien TT, Borand L, Quillet C, Connolly C, Lagarde D, Pym A, Lienhardt C, Dung NH, Taburet AM, Harries AD. Randomised pharmacokinetic trial of rifabutin with lopinavir/ritonavir-antiretroviral therapy in patients with HIV-associated tuberculosis in Vietnam. PLoS One. 2014 Jan 22;9(1):e84866. doi: 10.1371/journal.pone.0084866. eCollection 2014. PMID 24465443